CLINICAL TRIAL: NCT02504931
Title: SSRI Treatment of Dual Diagnosis PTSD and Alcohol Dependence: A Test of the Serotonergic Hypothesis
Brief Title: Serotonin Selective Reuptake Inhibitor Treatment of Dual Diagnosis Post-traumatic Stress Disorder and Alcohol Problems
Acronym: DDx
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: STRONG STAR Multidisciplinary PTSD Research Consortium (Unknown); South Texas Veterans Health Care System (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, John Roache, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: W81XWH0820117
Record Dates: First submitted 2013-07-16; First posted 2015-07-22 (Estimated); Results first posted 2018-02-27 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2017-04

CONDITIONS: PTSD; Alcohol Use Disorder
Keywords: PTSD; Alcohol; Dual Diagnosis; Sertraline; SSRI
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sertraline (Experimental): Subjects will receive a fixed dose of 150 mg sertraline per day. Sertraline dose will be gradually increased by giving sertraline subjects capsules filled with 50 mg for the first three days and then capsules filled with 100 mg for 4 days before beginning the 150 mg per day in the second week. After completing the study Visit 12, subjects will be given an additional two week supply of medicine to gradually taper down so as to minimize any withdrawal discomfort.
  Subjects in the Sertraline arm also will receive COPE therapy (Concurrent Treatment with Prolonged Exposure)which involves 12 sessions of manualized cognitive and behavioral therapy including exposure therapy for PTSD.
  Interventions: Drug: Sertraline
- Placebo (Placebo Comparator): Matching placebo capsules will be filled with corn starch only on the same schedule as the Sertraline.
  Subjects in the Placebo arm also will receive COPE therapy (Concurrent Treatment with Prolonged Exposure)which involves 12 sessions of manualized cognitive and behavioral therapy including exposure therapy for PTSD.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sertraline — A Randomized Controlled Trial Design will randomize subjects to one of two arms. Sertraline is the active medication treatment arm.
  Other Names: Zoloft
  Arms: Sertraline
Drug: Placebo — A Randomized Controlled Trial Design will randomize subjects to one of two arms. Placebo is the control medication treatment arm.
  Other Names: Placebo Control
  Arms: Placebo

SUMMARY:
The investigators propose to conduct a clinical trial to evaluate sertraline treatment efficacy in a large sample of military veterans with a dual diagnosis of PTSD and Alcohol Use Disorder who are receiving Cognitive and Behavioral Therapy as part of the VA-system's new dual diagnosis program. The study is designed as an efficacy trial of sertraline used as an adjunct to Cognitive Behavioral Therapy (CBT) in the treatment of PTSD/Alcohol dual diagnosis. There are two outcomes of interest, namely PTSD symptom improvement and also decreased alcohol consumption. The investigators are interested to know whether or not sertraline is superior to placebo in improving the symptoms of either one or both of these two disorders. Even though sertraline is a treatment of choice for PTSD, the investigators expect that the comorbid condition of alcohol dependence will complicate the treatment of PTSD and that the clustered subgroups will show differential treatment response with sertraline. The primary objective of the present study is to identify subgroups of alcohol dependent persons with PTSD who will either benefit or not benefit from treatment with SSRI's. The proposed study will enroll veterans with PTSD and dually-diagnosed alcohol dependence in a 12-week treatment providing sertraline vs. placebo medication as an adjunct to manualized CBT and will specifically test the hypothesis that subtypes of alcohol dependence can be used to predict which patients respond well and which subgroup responds poorly to SSRI treatment.

DETAILED DESCRIPTION:
Experimental Design. The study design is a parallel group, double-blind, placebo-controlled, stratified, randomized medication treatment trial of male and female veterans who experienced "in-theater" trauma and have both a PTSD and Alcohol Use dual diagnosis. All subjects will receive 12 weeks of manualized cognitive & behavioral therapy as a standard of care. Additionally, subjects will be randomized 1:1 to receive double-blind treatment with Sertraline vs. Placebo as an adjunctive treatment. The manualized therapy provides standard cognitive-behavioral therapy (CBT) addressing alcohol use and prolonged exposure (PE) behavioral therapy targeting PTSD. Sertraline is a common treatment for PTSD and psychiatric disturbance but is hypothesized to have differential efficacy in different subtypes of alcohol drinking patients. A stratified randomization scheme will balance placebo and sertraline assignment to two groups, and a post-hoc clustering approach will be used to determine which subgroups of dual diagnosis patients may benefit from sertraline vs. placebo treatment.

Veterans with PTSD who regularly drink more than 5 standard drinks of alcohol in a day (note one 12oz beer = one standard drink) may be eligible for the study if they meet criteria.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 year old Veterans with PTSD who regularly drink more than 5 standard drinks of alcohol in a day
* who experienced a trauma during deployment and
* who regularly drink more than 5 standard drinks alcohol and
* are interested in coming in once per week for 12 weeks of dual diagnosis individual therapy and
* are willing to participate in a placebo-controlled trial which could include receipt of sertraline (Zoloft).

Exclusion Criteria:

* if their PTSD Symptoms are adequately controlled by other medication regimens;
* they require inpatient alcohol detoxification; or currently receive naltrexone, disulfiram, acamprosate, or ondansetron treatment for alcohol dependence; or
* currently have an unstable medical illness; or
* have a bipolar or psychotic disorder; or
* currently are taking and are unwilling to discontinue taking any SSRI, SNRI, MAO inhibitor, tricyclic antidepressant, or anticonvulsant.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Roache, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- South Texas Veterans Health Care System, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sertraline: Subjects will receive a fixed dose of 150 mg sertraline per day. Sertraline dose will be gradually increased by giving sertraline subjects capsules filled with 50 mg for the first three days and then capsules filled with 100 mg for 4 days before beginning the 150 mg per day in the second week. After completing the study Visit 12, subjects will be given an additional two week supply of medicine to gradually taper down so as to minimize any withdrawal discomfort.
  Subjects in the Sertraline arm also will receive COPE therapy (Concurrent Treatment with Prolonged Exposure)which involves 12 sessions of manualized cognitive and behavioral therapy including exposure therapy for PTSD.
  Sertraline: A Randomized Controlled Trial Design will randomize subjects to one of two arms. Sertraline is the active medication treatment arm.
- Placebo: Matching placebo capsules will be filled with corn starch only on the same schedule as the Sertraline.
  Subjects in the Placebo arm also will receive COPE therapy (Concurrent Treatment with Prolonged Exposure)which involves 12 sessions of manualized cognitive and behavioral therapy including exposure therapy for PTSD.
  Placebo: A Randomized Controlled Trial Design will randomize subjects to one of two arms. Placebo is the control medication treatment arm.
Period: Overall Study
Arm/Group | Sertraline | Placebo
Started | 26 | 23
Completed | 14 | 13
Not Completed | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline | Placebo | Total
Number analyzed (Participants) | 26 | 23 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (13.4) | 41.2 (12.2) | 40.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 25 | 21 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 9 | 28
  Not Hispanic or Latino | 7 | 14 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 19 | 14 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 26 | 23 | 49
Region of Enrollment [Number; unit: participants]
  United States | 26 | 23 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percent Heavy Drinking Days
Description: Number of heavy drinking days in a 12 week period is reported by subjects and the percentage is calculated.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 26 | 23
percentage of days | 55.5 (24.8) | 65.1 (24.1)

2. Secondary Outcome: PTSD (Post Traumatic Stress Disorder) Symptom Score From PCL (Patient Monitoring Checklist)
Description: The PCL is a self-report measure that can be completed by patients in a waiting room prior to a session or by participants as part of a research study.
  The survey has 20 questions scored as:
  0=Not at all
  1. A little bit
  2. Moderately
  3. Quite a bit
  4. Extremely
  Interpretation of the PCL should be made by a clinician. The total symptom severity score is obtained by summing the scores for each of the 20 items to give a total of 1-80 points. The lower the score, the less severe the symptoms of PTSD, the higher the score, the more severe the symptoms.
Time Frame: 12 weeks of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sertraline | Placebo
Number analyzed (Participants) | 26 | 23
Units on a scale | 59.6 (9.6) | 61.7 (11.6)

ADVERSE EVENTS:
Time Frame: From baseline to 12 weeks.
Arm/Group | Sertraline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 23/26 | 18/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline (N=26) | Placebo (N=23)
Anxiety (Nervous system disorders) | 5 (5) | 2 (2)
Anger, hostility (Nervous system disorders) | 4 (4) | 0 (0)
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Depression (Nervous system disorders) | 5 (5) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 3 (3)
Drowsiness, dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Flu symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Insomnia (Nervous system disorders) | 6 (6) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4)
Nightmares (General disorders) | 5 (5) | 5 (5)
Pain (Nervous system disorders) | 8 (8) | 14 (14)
Difficulty concentrating (Nervous system disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (5) | 5 (5)
Headache (Nervous system disorders) | 8 (8) | 0 (0)
Irritability (Nervous system disorders) | 2 (2) | 0 (0)
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No